CLINICAL TRIAL: NCT05745116
Title: Evaluation of Repeated, In-Clinic, Self-Imaging by DME Patients Using the Notal Vision
Brief Title: Evaluation of Repeated, In-Clinic, Self-Imaging by DME Patients Using the Notal Vision Home OCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2022.001
Record Dates: First submitted 2023-01-06; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Notal Vision Home OCT — Optical Coherence Tomography (OCT) was originally developed in 1991 as a non-invasive imaging technology to generate cross-sectional imagery of ocular tissues in vivo1. Cross-sectional visualization of the retina has proven to be a valuable tool in the identification and assessment of structural abnormalities that are not visible with ophthalmoscopic or biomicroscopic examination. OCT has become eye care professionals' leading diagnostic tool in the detection, diagnosis and treatment of retinal diseases and conditions, including age-related macular degeneration (AMD), Diabetic Macular Edema (DME), and Retina Vein Occlusion (RVO). Notal Vision, Inc. (Manassas, VA) is developing a Home Optical Coherence Tomography (OCT) System to allow OCT images to be captured on an OCT device placed in the patients' homes for daily scanning of eyes diagnosed with DME. This Home OCT allows visualization of retinal fluid in the central 10 degrees and is currently for investigational use only.

SUMMARY:
Evaluation of Repeated, In-Clinic, Self-Imaging by DME Patients Using the Notal Vision Home OCT The purpose of this study is to collect data on the NVHO device at up to three sites.

DETAILED DESCRIPTION:
7 Study Procedures and Office Visit Schedule Informed Consent Voluntary informed consent will be obtained from every subject prior to the initiation of any screening or other study related procedures. The Investigator must have a defined process for obtaining informed consent. Specifically, the Investigator, or designee, will explain the clinical study to each potential patient and the patient must indicate voluntary consent by signing and dating of the approved informed consent form. The patient must be provided an opportunity to ask questions to the Investigator, and if required by local regulation, other qualified personnel.

Description of Study Procedures and Visits 7.2.1 Office Visit NOTE: Any planned treatment for DME at the day of the study should be administered after completion of all study-related scans

At the enrollment Office Visit, the exams will be conducted in the following order:

1. Patient will be informed concerning the study and sign the Informed Consent Form (ICF) prior to conduct of any study procedures. 2. Following signing the ICF, subjects will be assigned a Subject ID by a designated staff at the clinical site. 3. The following data will be collected for each study subject:

1. Date of birth
2. Gender
3. Number and type of Anti-VEGF injections and last injection date 3. Refraction correction 4. Snellen BCVA on both eyes on the day of the visit. 5. Eligible eye(s) of the subject will be scanned, non-dilated, with a Zeiss Cirrus or Spectralis OCT device with one (1) acceptable volume scan of each eye being obtained out of up to 3 attempts.

Scanning pattern to be used:

Zeiss Cirrus: Macular cube, 6X6mm, 128 B-scans per volume scan Or Spectralis: "Dense" preset (scan size: 20°x20°, # section images: 49, # ART Mean: 16, scan angle cSLO image: 30°, image resolution: High speed) centered on the fovea.

R&D DOCUMENTS C2022.001 Subject: Single In-Clinic Encounter with the Notal Vision Home OCT Page: 11 OF 18 Version 3 FOR CONFIDENTIAL USE ONLY October 2022 6. Eyes of the subject that meet all screening criteria will be enrolled. If both eyes of the subjects meet all screening criteria both eyes will be enrolled. NOTE: Approximately 90% of the enrolled subjects should have at least one eye with DME at the time of enrollment. 7. The following data will be collected for the study eye(s):

a. Qualifying diagnosis for the study eye from the subject's medical record b. From the subject's medical record, the presence of other ophthalmic conditions including but not limited to: i. Cataract ii. Glaucoma iii. Dry Eye iv. Other macula findings, e.g., epi retinal membrane, macular hole, vitreo-macular traction (VMT) Following confirmation of subject eligibility, subject will be placed in a room with the NVHO device which has been set up by a technician.

1. The technician will register the subject using the touchscreen of the NVHO device.
2. The subject will perform a self-tutorial. The training flow begins with demonstration clips followed by a practice session. The training flow will be followed by a self-scan that the system uses as a calibration session.
3. Following completion of the training, the clinic technician shall set the device for selfscanning flow.
4. Following the training, the subject must complete a unsupervised successful calibration scan on each study eyes. The technician will check the status of the calibration scan (success/failure) using a dedicated screen on the device, presented at the end of each scanning session. Each study eye has up to 3 attempts to complete a successful calibration scan.
5. If an eye went through a successful calibration scan, a "Success" message, in green letters, will be presented on the dedicated screen, at the end of the session and this eye will be ready to start the scanning phase.
6. In case of failure in all 3 calibration attempts, an error message "3 successive calibrations failed" will be presented in red letters on the dedicated screen. In that case this eye should be excluded from the study and the technician should prevent the patient from re-scanning it. R&D DOCUMENTS C2022.001 Subject: Single In-Clinic Encounter with the Notal Vision Home OCT Page: 12 OF 18 Version 3 FOR CONFIDENTIAL USE ONLY October 2022
7. Scanning phase - the subject will perform four (4) unsupervised self-scans on each study eye with a rest period of ~2 minutes between self-scans.

5. AEs, if applicable, will be collected. 6. Exit subject from the study 7. Self-scan data will be backed up on the NVHO device. 8. Study visit data will be registered into the sponsor-provided CRF and sent to Notal The Zeiss Cirrus or Spectralis OCT images will undergo anonymization process using identical CRF name and number of the subject and will be sent to Notal. Discontinued Subjects Discontinued subjects are those who withdraw or are withdrawn from the study after being successfully consented into the study. Subjects may discontinue from the study at any time for any reason. Subjects may be discontinued from the study at any time if, in the opinion of the Investigator, their continued participation poses a risk to their health. Discontinued subjects will not be replaced (i.e., their subject number will not be reassigned or reused.) An Exit form must be completed for all subjects. Clinical Study Initiation and Termination Before the study can commence, the Sponsor or its designee must ensure that all relevant study documents are available and that the Site Initiation has been performed. Only then can arrangements be made for start of recruitment. If the clinical study is terminated or suspended, the Sponsor will inform the Investigator and the regulatory authorities of the termination/suspension and the reasons for the termination/suspension.

The Investigator should promptly notify the IEC/IRB (Independent Ethics Committee/Institutional Review Board) of the termination/suspension and of the reasons. The Sponsor reserves the right to close the investigational site or terminate the study in its entirely at any time, for reasonable cause.

Reasons for the closure of an investigational site or termination of a study may include:

1. Successful completion of the study
2. Study enrollment goals are met
3. Investigator fails to comply with the protocol or GCP guidelines
4. Safety concerns
5. Sufficient data suggesting lack of efficacy
6. Inadequate recruitment of patients by the Investigator The investigator also may terminate the study at his/her site for reasonable cause. If the Sponsor terminates the study for safety reasons, it will immediately notify the Investigator by telephone and subsequently will provide written confirmation and instructions for study termination.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak, read and understand English.
* Ability to agree, understand and sign the informed consent form.
* Eighteen (18) years of age or older at the time of Informed Consent.
* Subjects diagnosed with DR (Diabetic Retinopathy) in at least one eye, with or without DME
* Best corrected Visual Acuity of 20/320 (6/96) or better in eyes participating at the study.

Exclusion Criteria:

* Subjects with dilated pupils.
* Subjects with other retinal disease requiring steroidal or anti-VEGF injections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include up to one hundred fifty (150) patients, with DR in at least one eye at the time of enrollment. Subjects will be enrolled at up to three (3) sites in the United States.
  The subjects must meet all inclusion / exclusion criteria. Approximately 90% of the enrolled subjects should have at least one eye with DME at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate subjects' ability to perform multiple OCT self-scanning following a self-tutorial on the Notal Vision Home OCT (NVHO) | within 2 hours of an office visit
  % of completion a self-imaging session
Evaluate the repeatability of the Notal OCT Analyzer (NOA) automatic fluid volume quantification in volume scan from self-scanning with the NVHO in the central 10 degrees of the macula of Diabetic Retinopathy (DR) patients | within 2 hours of an office visit
  NVHO volume scan Total Retinal Fluid (TRF) amount measured by NOA, NVHO volume scan Intra-Retinal Fluid (IRF) amount measured by NOA, NVHO volume scan Sub-Retinal Fluid (SRF) amount measured by NOA
Compare fluid quantification in images from NVHO and a commercial OCT | within 2 hours of an office visit
  Compare fluid quantification in images captured by the NVHO, as calculated by the Notal OCT Analyzer (NOA) algorithm and the fluid quantification in images captured by a commercial OCT, as marked by a human reader - in the central 10 degrees of the macula of DR patients Zeiss Cirrus or Spectralis OCT volume scan Total Retinal Fluid (TRF), Intra-Retinal Fluid (IRF), Sub-Retinal Fluid (SRF) amount measured by a human reader
Scanning session completion status - complete/incomplete | within 2 hours of an office visit

SECONDARY OUTCOMES:
Safety Endpoints | within 2 hours of an office visit
  All adverse events (AEs) occurring during the conduct of this study will be captured and reported.
  All exam procedures will be conducted as a part of the subject's routine care. While it is unlikely that an adverse event will occur, all events will be reported.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Elman Retina Group, PA, Baltimore, Maryland
  - The Retina Group of Washington, Fairfax, Virginia
  - Wagner Kapoor Research Institute, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided